CLINICAL TRIAL: NCT05996614
Title: Evaluation of Platelet Rich Plasma in Skin Graft Take for Patients With Post Burn Raw Areas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ibrahim Ragab Ibrahim ali, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRP in skin grafts
Record Dates: First submitted 2022-10-07; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Skin Burn
MeSH Terms: conditions — Paresthesia | interventions — Skin Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group with PRP (Experimental): Group of patients with post burn raw areas treated with application of platelet rich plasma
  Interventions: Procedure: PRP in skin grafts
- group without PRP (Experimental): Group of patients with post burn raw areas treated with conventional methods
  Interventions: Procedure: conventional methods in skin grafts

INTERVENTIONS:
Procedure: PRP in skin grafts — topical application of platelet rich plasma before resurfacing with STSG in Post burn raw areas
  Arms: group with PRP
Procedure: conventional methods in skin grafts — fixation of the graft with stitches and staplers
  Arms: group without PRP

SUMMARY:
1. To evaluate the effect of the platelet rich plasma on the take of split thickness skin graft and its early and late results in resurfacing of post burn raw areas.
2. To evaluate the effect of PRP on wound healing on skin graft donor site.

DETAILED DESCRIPTION:
Burn injuries involve tissue destruction due to energy transfer,The burn injuries can be caused by heat from hot liquids, solids or fire, an less common causes are friction, heat, chemical or electric sources The treatment of burns is complex due to the combination of hypermetabolic physiological response and the need for good functional and cosmetic recovery. Split thickness skin grafts (STSGs) are commonly used to resurface large areas of Post burn raw areas.

The time to complete wound healing ranged from 2 to 75 days. Factors that significantly affected time to complete wound healing were graft loss by seroma, presence of hypergranulation tissue, premorbid conditions, and total body surface area burned.

Generally, skin graft undertakes three steps for healing: anchorage, inosculation, and maturation. Haematoma, shearing, and infection on recipient sites of skin graft can reduce skin graft take, and even lead to skin graft loss.

Platelet-rich plasma (PRP) is an autologous blood-derived biomaterial that is enriched with a 2- to 6-fold concentration of platelets in comparison to normal human platelet concentration. Multiple growth factors and bioactive proteins are stored in α-granules of platelets. These growth factors can promote proliferation of endothelial cells, epithelial cells as well as fibroblasts, and increase angiogenesis. The potential clinical application of PRP in skin graft might rely on its haemostasis, adhesive, antibacterial and healing properties.

ELIGIBILITY:
Inclusion Criteria:

1. Age (15- 60 years).
2. Post burn Raw area less than 10 % of total body surface area .
3. Selected donor sites.

Exclusion Criteria:

1. Raw area due to other causes ( trauma, ischemia,..etc)
2. Patients with bleeding tendency.
3. Patients with comorbidities(diabetes, malignancy,..etc)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
histopathological biopsy from both groups by punch Biopsy (vancouver scale ) | 3 months
  pigmentation (0-2) ,normal 0, Hypopigmentation 1 ,Hyperpigmentation 2 Vascularity (0-3) ,Normal 0, Pink 1, Red 2, Purple 3 Pliability (0-5) Normal 0 ,Supple 1 ,Yielding 2,Firm 3, Banding 4, Contracture 5 Height (0-3) Normal(flat)0 ,(0-2mm)1,(2-5mm)2,(>5mm)3

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Elsonbaty, prof, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia-Sanchez JM, Mirabet Lis V, Ruiz-Valls A, Perez-Plaza A, Sepulveda Sanchis P, Perez-Del-Caz MD. Platelet rich plasma and plasma rich in growth factors for split-thickness skin graft donor site treatment in the burn patient setting: A randomized clinical trial. Burns. 2022 Nov;48(7):1662-1670. doi: 10.1016/j.burns.2021.10.001. Epub 2021 Oct 22. PMID 34952738